CLINICAL TRIAL: NCT00830505
Title: A Randomized, Double-Blind, Cross-Over Study to Demonstrate Superiority of Fluticasone/Salmeterol Over Double the Dose of Fluticasone on Methacholine Hyper-Reactivity in Patients With Persistent, Mild to Moderate Asthma
Brief Title: Fluticasone/Salmeterol (FP/SM) Versus Double the Dose Fluticasone (FP) in Patients With Mild to Moderate Asthma
Acronym: CLE001
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLE001
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Asthma
Keywords: fluticasone; salmeterol; bronchoprotection
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1: fluticasone/salmeterol (Experimental): 2 puffs twice a day for 2 weeks
  Interventions: Drug: fluticasone/salmeterol
- 2: fluticasone (Active Comparator): 2 puffs twice a day for 2 weeks
  Interventions: Drug: fluticasone

INTERVENTIONS:
Drug: fluticasone/salmeterol — 2 puffs twice a day for 2 weeks
  Other Names: fluticasone/salmeterol combination
  Arms: 1: fluticasone/salmeterol
Drug: fluticasone — 2 puffs twice a day for 2 weeks
  Other Names: Flixotide
  Arms: 2: fluticasone

SUMMARY:
The purpose of this study is to compare the effects of Fluticasone/ salmeterol combination and double the dose of fluticasone on airway hyper-responsiveness to methacholine in a randomised, double blind, double dummy, cross-over trial.

DETAILED DESCRIPTION:
The objective of pharmacotherapy in the treatment of asthma is restoration of pulmonary function. This is accomplished by reducing airway inflammation, stimulating bronchodilation or a combination of the two. The classes of drug that have proved effective in this regard are anti-inflammatory agents such as corticosteroids and mast cell-stabilising agents, and bronchodilators such as β2 adrenergic agonists.

Inhaled corticosteroids (ICS) are used as a first-line anti-inflammatory prophylactic therapy for asthma. Current guidelines recommend initiating treatment with a medium to high dose, then reducing to the lowest effective dose for long-term maintenance.

Corticosteroids are preferably inhaled from aerosol inhalers (commonly pMDIs: pressurised metered dose inhalers) using large-volume spacer devices for pMDI doses in excess of 800 µg/day of BDP (Beclometasone Dipropionate), or equivalent. CFCs ((Chlorofluorocarbon)) ( propellants in BDP pMDIs are being replaced with non-ozone-depleting propellants such as hydrofluoroalkane-134a (HFA).

Comparison of steroid therapies in patients with asthma is rather difficult using conventional measures such as lung function parameters (FEV1/forced expiratory flow over one sencond or PEF/Peak expiratory flow) when chosen as the primary outcome variable, as these are relatively insensitive to ICS therapy, and are rather distant from the underlying inflammatory process. Measurements of airway responsiveness are frequently used to evaluate asthma treatments and methacholine or histamine challenge testing is recognized and recommended by regulatory authorities.

Airway responsiveness is defined as the relative ease with which airways can be made to constrict when exposed to non-sensitising chemical or physical stimuli such as methacholine, histamine, cold air, exercise or hyperventilation. Methacholine challenge looks at the functional antagonism of long acting bronchodilators (LABA) against increased airway tone; as such there is always more room for potential improvement, and therefore treatment response, with protection against challenge than with spirometry alone. In addition the effect of ICS is more sensitive when measured with methacholine challenge testing than with lung function alone.

In this study, which looked at the effect of both ICS alone and ICS with LABA, methacholine challenge was selected as it is more sensitive than lung function alone.

The methacholine challenge test involves delivering doubling concentrations of methacholine over a period of time (usually 2 minutes) until a given level of bronchoconstriction is achieved (often a 20% fall in FEV1). The provocative concentration producing a 20% fall in FEV1 is termed the PC20. Previous studies have shown that treatment with 50µg salmeterol versus 100 µg Fluticasone plus 50 µg salbutamol showed a 1.15 doubling dose difference in response to methacholine challenge, which would indicate that a treatment response to the 100µg fluticasone would be in the region of 1 doubling dose15. A similar study demonstrated a similar (0.9 dd difference between treatments) when comparing FPSM/fluticasone/ salmeterol (125/50µg) vs FP/Flutiocasone Propionate(250µg) alone.

One doubling dose can therefore be shown to indicate a clinically relevant difference between the treatments (based upon either the ICS or the LABA component of the combination product) as shown in previous studies. Therefore 1 dd shift in treatment response was defined as the minimally important clinical difference for the purposes of the statistical calculations.

In addition to the measures of efficacy, this study aimed to compare the effect of the two treatments on basal HPA-axis suppression in vivo, as measured by the ratio of overnight urinary cortisol to creatinine.

The bioactivity of a corticosteroid is thought to be related to the relative degree of HPA-axis suppression as measured by the decrease in the ratio of overnight urinary cortisol to creatinine. This measure has been shown to be as sensitive as a 24-hour collection. An alternative, though less sensitive, assessment is plasma cortisol and creatinine production 30 minutes after stimulation with ACTH19,20.

The two formulations were administered for 2 weeks, which was thought to be sufficient to achieve steady state in terms of HPA-axis suppression. It had been shown previously that steady state plasma levels can be achieved in 3 days when using fluticasone propionate.

Smokers have been shown to develop acquired steroid resistance, resulting in a diminished response. It has therefore been the practice of most studies on asthma to exclude smokers as a matter of course. Indeed current asthma guidelines are based on these studies. A recent subgroup analysis of the 'Gaining Optimal Asthma controL (GOAL) study' reported by Pedersen and colleagues has revealed some interesting results. They discovered that smokers gained more benefit from FPSM vs FP alone, as compared to non smokers, in terms of reduction in exacerbation rates over 12 months.

To put the results of this study into a clinical context, in the majority of patients who were non smokers it would take 25 years to obtain an additional benefit to prevent an exacerbation by taking fluticasone/salmeterol vs fluticasone alone. In smokers it would take 6.66 years to see the same benefit conferred by using combination therapy.

The reasons for the apparent increased benefits of treatment with FP/SM in smokers are unclear. A potential explanation for this could be that, in the face of the relative steroid resistance seen in smokers, the smooth muscle stabilisation conferred by the LABA becomes of greater significance. Another possible explanation is that smoking induces greater hyper-reactivity in the airway smooth muscle, which responds well to the smooth muscle stabilisation offered by LABAs. A third possibility is that smoking might in some way up-regulate beta2- adrenoreceptor function. It was therefore felt important to include a cohort of smokers in this study.

To enter Treatment Period 1, subjects must have had a provocative concentration of methacholine causing a 20% decrease in FEV1 (PC20) of less than 4mg/mL at randomisation and FEV1 at the end of the run-in period and wash-out must have remained within 15% of that recorded at screening, and ≥ 60% predicted.

For entry into the second treatment period the PC20 after 2 to 3 weeks of the placebo washout must have been within ±1 doubling dilution of the initial placebo run in period.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent given by patient.
2. Male or female patients between 18 and 65 years of age inclusive.
3. Persistent stable asthmatics (FEV1 > 60%)
4. On ≤ 1000 µg FP or equivalent or if on combination therapy up to 500 µg of FP or equivalent (e.g. FP/SM 125 2-puffs BD or BUD/FM 200/6 2-puffs BD)
5. Patients suffering from stable, persistent, mild to moderate asthma as defined by GINA Guidelines and for whom FEV1 > 60 %
6. In the opinion of the investigator, able and willing to comply with the requirements of the protocol.

Exclusion Criteria:

1. Severe asthmatics as defined by an FEV1 < 60% or PEF variability >30% or with continual daytime or nocturnal symptoms.
2. Known or suspected hypersensitivity to FP or any other constituents of the Test or Reference pMDI
3. Any clinically significant medical condition or abnormality, which, in the opinion of the investigator, might compromise the safety of the patient or which might interfere with the study (such as unstable angina, acute myocardial infarction in the preceding 3 months, recent TIA / CVA).
4. Females who are pregnant, lactating or planning to become pregnant.
5. Approximately half of the subjects will be smokers and half currently non-smokers (or who have ceased smoking at least 1 year previously).
6. Clinically significant laboratory values, as judged by the investigator.
7. Receipt of an investigational drug within 30 days or 5 half-lives, whichever is longer, prior to the screening visit.
8. Patients who are scheduled to receive any other investigational drug during the course of the study.
9. Concomitant use of medicines (prescribed, over the counter or herbal) that may interfere with the trial.
10. Exacerbations of asthma requiring oral steroids, hospitalisation or change in asthma therapy in the previous three months.
11. Respiratory tract infection in the previous 2 months.
12. Patients with significant concomitant respiratory disease such as COPD, CF, ABPA, active pulmonary TB or bronchiectesis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
methacholine challenge | before and after a 2 week treatment period
  methacholine challenge

CONTACTS AND LOCATIONS:
Overall Officials: Karine L Clearie, MBBS, MRCP, Principal Investigator — Asthma and Allergy Research Group; Brian J Lipworth, MBchB, Study Director — Asthma and Allergy Research Group
Locations (1):
- Asthma and Allergy Research Group, Dundee, Angus, United Kingdom

REFERENCES:
- [Result] Clearie KL, McKinlay L, Williamson PA, Lipworth BJ. Fluticasone/Salmeterol combination confers benefits in people with asthma who smoke. Chest. 2012 Feb;141(2):330-338. doi: 10.1378/chest.11-0392. Epub 2011 Jun 2. PMID 21636667
- See also: Chest. 2012 Feb;141(2):330-338. doi: 10.1378/chest.11-0392. Epub 2011 Jun 2. — http://doi.org/10.1378/chest.11-0392